CLINICAL TRIAL: NCT00556647
Title: A Prospective, Open, Single Center, Study of One-day Diagnostic Track for Lung Cancer Suspects From Chest X-ray Using PET-CT and Subsequent Multiple Endoscopic Investigations. (Including Bronchoscopy, EUS-FNA)
Brief Title: Fast-track Diagnosis for Lung Cancer Suspects With PET-CT and EUS
Status: Completed | Type: Observational
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Jan W.K. van den Berg, Dr., Isala
Other Study IDs: NL12541.075.06
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Lung Cancer
Keywords: fast-track diagnosis; PET-CT; endoscopic techniques; lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: Fast-track diagnosis
  Interventions: Procedure: fast track diagnosis; Procedure: conventional diagnosis

INTERVENTIONS:
Procedure: fast track diagnosis — fast-track diagnosis, PET-CT, bronchoscopy
Procedure: conventional diagnosis — out-patient diagnosis

SUMMARY:
Patients who are admitted to the outpatient pulmonology department by a general practitioner or specialist with a chest X-ray suspicious for lung cancer with an age between 18 and 80 years are suitable for participation. The X-ray and referral are studied by a chest physician (by phone or fax ). Selected patients are invited to enter the study after answering a questionnaire by phone (p. 31). The questionnaire screens patients' interest, co-morbidity and medication use. Informed consent forms, patient information forms and a time table for the diagnostic day are provided by mail or E-mail in cases where time gets short. Waiting time to enter the study will be no longer than one week.

Hundred patients will be recruited by means of informed consent. Patients will be admitted at the pulmonary ward for the study day and will be accompanied by nurses. All patients will get PET-CT scanning in the morning of the study day. Depending on the location of lesions seen on PET-CT, further invasive diagnostic procedures will be planned for the afternoon.

Mediastinal and adjacent structures will be analysed with EUS-FNA. Mediastinal staging will be done with bronchoscopy alone for central located tumors, peripherally located lesions will be analysed with EUS-FNA or bronchoscopy.

The percentage of patients in which this diagnostic track leads to a diagnosis and tumor stage in one day will be determined. The number of tests and diagnostic procedures needed to obtain a diagnosis, including tumor stage (especially final stage NSCLC) and function tests, will be compared with a historical matched study group. This historical study group is chosen from an era before the availability of integrated PET-CT and ultrasound guided endoscopic tools and meets the same inclusion and exclusion criteria as the patients in this study. The timelines from initial chest X-ray to diagnostic day to informing the patient to start of treatment will be determined. These figures will be compared with the historical study group.

DETAILED DESCRIPTION:
Background of the study:

Patients have to pass different diagnostic phases in their analysis of a chest X-ray suspicious for lung cancer. Long waiting times with uncertainty about the outcome are a waste of time and unacceptable for the patient. Hospital visits as a consequence of this are a financial burden. Important reasons for physicians to shorten diagnostic tumor analysis. Shortening and intensifying the diagnostic track by combining diagnostic and staging procedures would preclude unnecessary tests and procedures, lowering the total hospital costs per patient and may lead to more satisfaction for patient and physician.

PET-CT is the most important imaging tool for lung cancer analysis and better than CT or FDG-PET alone, but not optimal for determination of tumour invasion in mediastinal or other adjacent structures. MRI is more suitable for this purpose, but is limited available. EUS-FNA (carinal lymph nodes), eventually in combination with CT or FDG-PET and EBUS-TBNA (right mediastinal lymph nodes), superior to TBNA alone, are novel imaging techniques with a high accuracy. Bronchoscopy provides information on tumour type and resectability of centrally but not peripherally located tumours. Mediastinal staging can be performed by adding TBNA to bronchoscopy with high accuracy. PET-CT, as a superior imaging mode, could direct for the best subsequent endoscopic technique for obtaining a tissue diagnosis as well as leading to a more comprehensive staging of patients with suspected lung cancer.

False negative findings could be caused by sampling errors or false interpretations by the cytopathologist of specimens with tumour cell poverty. A more sensitive immune histochemical analysis could modify EUS-FNA and EBUS-TBNA results.

Objective of the study:

1. to study feasibility of a fast one-day diagnostic track including PET-CT and subsequent diagnostic/ staging investigation depending on PET-CT findings.

   to determine:
2. the percentage of patients in which the one-day track is sufficient for diagnosis and staging needing no more further investigations.
3. the time-spans needed for diagnosis (including staging and function tests) of the patients in comparison to a historical study group.
4. the amount of investigations needed to obtain the diagnosis compared with a historical study group.
5. the effect of immuno-histochemical analysis on the sensitivity of data of diagnostic procedures.

Study design:

A Prospective, open, single center, study.

Patients who are admitted to the outpatient pulmonology department by a general practitioner or specialist with a chest X-ray suspicious for lung cancer with an age between 18 and 80 years are suitable for participation. The X-ray and referral are studied by a chest physician (by phone or fax ). Selected patients are invited to enter the study after answering a questionnaire by phone ( p. 31).

The questionnaire screens patients' interest, co-morbidity and medication use. Informed consent forms, patient information forms and a time table for the diagnostic day are provided by mail or E-mail in cases where time gets short. Waiting time to enter the study will be no longer than one week.

Hundred patients will be recruited by means of informed consent. In a narrow logistic scheme the study subjects will undergo a diagnostic work up to a maximum of 3 patients per study day (p. 32). Patients will be admitted at the pulmonary ward for the study day and will be accompanied by nurses. All patients will get PET-CT scanning in the morning of the study day. Depending on the location of lesions seen on PET-CT, further invasive diagnostic procedures will be planned for the afternoon, according to a scheme outlined on page 33. In the meanwhile, routine blood tests, EKG and pulmonary function tests are done. The invasive diagnostic procedure to be chosen, has to provide ideally a diagnosis and stage at one time.

Mediastinal and adjacent structures will be analysed with EUS-FNA or EBUS-TBNA. EBUS-TBNA will be used for right mediastinal lymph nodes. Carinal lymph nodes are biopsied with EUS-FNA. Mediastinal staging will be done with bronchoscopy alone for central located tumors, peripherally located lesions will be analysed with EUS-FNA or bronchoscopy in combination with EBUS-TBNA.

When enough material is available, cytologic specimen will be stored in cell casts fixed in agar. In case of negative biopsies, surgical verification follows. When this verification proves that cytologic biopsies were false negative, immune histochemical analysis on the agar imbedded material will be done retrospectively.

When patients are recovered from their diagnostic procedure, they will leave the hospital with an appointment for a visit one week later to be informed about their diagnosis and treatment. Additive appointments will be made on a term as short as possible and necessary when extra diagnostic tests are needed like MRI, exercise tests, perfusion tests or evaluation by other consultants.

The percentage of patients in which this diagnostic track leads to a diagnosis and tumor stage in one day will be determined. The number of tests and diagnostic procedures needed to obtain a diagnosis, including tumor stage (especially final stage NSCLC) and function tests, will be compared with a historical matched study group. This historical study group is chosen from an era before the availability of integrated PET-CT and ultrasound guided endoscopic tools and meets the same inclusion and exclusion criteria as the patients in this study. The timelines from initial chest X-ray to diagnostic day to informing the patient to start of treatment will be determined. These figures will be compared with the historical study group.

Finally, patients will be asked to fill in a patient satisfaction questionnaire concerning the one-day diagnostic program track, the informative visit and after an eventual successive treatment start (p. 31).

Study population:

Hundred patients with suspicion of lung cancer on X ray with an age between 18-85 years admitted to the pulmonologist by their general practitioner or specialist.

Intervention (if applicable):

One-day diagnostic track using PET-CT eventually with bronchoscopy, EUS-FNA , EBUS-TBNA and ultrasound guided transcutaneous biopsies.

Primary study parameters/outcome of the study:

1. Number of patients that will have a definitive diagnosis and final stage NSCLC in one day.
2. Time between chest X-ray with suspicion on lung cancer and the first visit to the outpatient clinic.
3. Time between the first outpatient clinical contact and informing patient about definite diagnosis.
4. Time from the definite diagnosis until the initiation of therapy.

Secundary study parameters/outcome of the study (if applicable):

1. Number of patients able to have all diagnostic tests in one-day.
2. Number of tests and procedures that have been performed.
3. Patient satisfaction with the one-day procedure.
4. Sensitivity of EUS-FNA and EBUS-TBNA when immunohistochemical analysis is added to investigate false negative procedures.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness (if applicable):

There are no different adverse effects due to the diagnostic program. Patients in the one-day diagnostic track will undergo the same diagnostic interventions as patients outside the study. The risk of bleeding and infection due to the EUS and EBUS procedures must be mentioned, although patients would be undergo these biopsies even if they would not participate to this trial; there is no 'additive risk'.

The burden is that the whole diagnostic program could lead to psychological distress because of the several investigations within a relatively short period. Patients with claustrophobia might be anxious during the PET-CT. The expected benefits are a patient satisfaction due to short diagnostic timeframes, lesser diagnostic procedures and faster decision making in therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

* patients with a suspicion of lung cancer on chest X-ray
* age between 18-85 years
* informed consent.

Exclusion Criteria:

* comorbidity (alcoholabuse, drugsabuse and limiting psychiatric disease)
* non-compliance
* previous diagnostic tests for the suspicious X-ray (endoscopy, CT)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected of lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2006-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Number of patients that will have a definitive diagnosis and final stage NSCLC in one day | 1 day

SECONDARY OUTCOMES:
Number of tests and procedures that have been performed. Patient satisfaction with the one-day procedure. Sensitivity of EUS-FNA and EBUS-TBNA when immunohistochemical analysis is added to investigate false negative procedures. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: J. Stigt, Drs., Study Director — Isala
Locations (1):
- Isala Klinieken, Zwolle, Netherlands